CLINICAL TRIAL: NCT04548206
Title: Effect of Pilates Training on Sensory, Muscle Strength, Balance, and Gait in Patients With Multiple Sclerosis
Brief Title: Effect of Pilates Training in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Cagla Ozkul, Research Assistant, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 166
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; sensation; gait; Pilates
MeSH Terms: conditions — Multiple Sclerosis | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: prospective randomize controlled study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates training (Experimental): 60 minutes of Pilates training will be performed for 8 weeks.
  Interventions: Other: Pilates training
- Control group (Placebo Comparator): The control group will be taught relaxation exercises and will be asked to perform the exercises at home.
  Interventions: Other: control

INTERVENTIONS:
Other: Pilates training — The program consisted of core-based Pilates exercises on the mat for 60 minutes.
  Arms: Pilates training
Other: control — The program consisted of progressive relaxation exercises at home.
  Arms: Control group

SUMMARY:
Knee flexor and extensor muscle weakness in MS patients causes a decrease in walking distance and is an important determinant of walking capacity. Exercise training has beneficial effects on muscle strength, balance, and walking in MS patients. Although the effects of aerobic and resistant exercise training in MS patients are often emphasized, today the effect of different exercise types is also wondered. Pilates is a core stability-based exercise method that improves endurance, flexibility, movement, posture, and respiratory control. The aim of this study is to examine the effect of Pilates training on sensation, muscle strength, balance, and walking in MS patients.

DETAILED DESCRIPTION:
Patients with MS between 0-5,5 score according to the Extended Disability Status Scale (EDSS) will be included in the study. The balance, gait, position sense, and muscle strength will be evaluated. The study was designed as a prospective, randomized controlled study. The patients will be randomly assigned to two groups, the "Pilates training" group, and the control group. Pilates training will be performed by the Pilates training group 2 times for 8 weeks under supervision in the outpatient clinic. The control group will be taught relaxation exercises and will be asked to perform the exercises 2 times for 8 weeks at home. Statistical analyses will be performed using the SPSS software version 15 (SPSS Inc. Chicago, IL, USA). The pre-training and post-training measurements of groups will be compared with the paired sample t-test.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Having a diagnosis of "Multiple Sclerosis"
* Relapse free in the last 3 mounts
* Having an ambulatory status (Expanded Disability Status Scale score ≤ 6 )
* No diagnosis of depression

Exclusion Criteria:

* Any cardiovascular, orthopedic, visual, hearing and perception problems that may affect the results of the research.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Gait | 5 minutes
  Gait parameters will be assessed via the G-Walk on two separate occasions. The G-Walk is a device that is worn on the waist via an elastic belt. The G-Walk is built with a triaxial accelerometer 16 bit/axes with multiple sensitivity, a triaxial magnetometer 13 bit and a triaxial gyroscope 16 bit/axes with multiple sensitivity. This hardware is capable of acquiring and transmitting data to a computer through a Bluetooth connection and at the end of each analysis an automatic report containing the gait assessment results is ready to be analyzed.
  Gait symmetry values of the right and left sides are obtained within this report. While the symmetry index ranges from 0 to 100, a value closer to 100 indicates that the gait is more symmetrica.
Balance | 10 minutes
  The Modified Sensory Organization Test, which is performed using computerized posturography, measures postural sway in response to 4 different sensory conditions is measured using a force platform.
Light touch-pressure sensation | 10 minutes
  Light touch-pressure sensation will be assessed using a full Semmes-Weinstein Monofilament (SWM) test kit (North Coast Medical, San Jose, CA, USA).
Vibration sensation | 10 minutes
  Duration of vibration sensation will be measured using 128-Hz frequency tuning fork (Elcon1 Medical Instruments, Tuttlingen, Germany).
Two-point discrimination | 10 minutes
  Two-point discrimination sensation of the foot sole will be evaluated using an aesthesiometer (Baseline1, White Plains, New York, USA).
Position sensation of knee joint | 5 minutes
  Open kinetic chain position of both knees will be evaluated using a Dualer IQ Digital Inclinometer (J-Tech Medical, Midvale, UT, USA).
Knee proprioception | 10 minutes
  Knee proprioception will be evaluated with the active joint reposition test using the isokinetic system (Cybex Norm, Humac, CA, USA).
Position sensation of trunk | 10 minutes
  Position sensation of trunk will be evaluated using a Dualer IQ Digital Inclinometer (J-Tech Medical, Midvale, UT, USA).
Knee strength | 20 minutes
  Knee strength will be evaluated using the isokinetic system (Cybex Norm, Humac, CA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Cagla Ozkul, Phd, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citaker S, Gunduz AG, Guclu MB, Nazliel B, Irkec C, Kaya D. Relationship between foot sensation and standing balance in patients with multiple sclerosis. Gait Posture. 2011 Jun;34(2):275-8. doi: 10.1016/j.gaitpost.2011.05.015. Epub 2011 Jun 16. PMID 21683600
- [Background] Bulguroglu I, Guclu-Gunduz A, Yazici G, Ozkul C, Irkec C, Nazliel B, Batur-Caglayan HZ. The effects of Mat Pilates and Reformer Pilates in patients with Multiple Sclerosis: A randomized controlled study. NeuroRehabilitation. 2017;41(2):413-422. doi: 10.3233/NRE-162121. PMID 28946576